CLINICAL TRIAL: NCT00708877
Title: Liver Transplantation for Cholangiocarcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: study procedures have become standard of care as patients seeking Model for End-Stage Liver Disease (MELD) exception points for cholangiocarcinoma
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI18450
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Results first posted 2012-04-04 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Cancer; Cholangiocarcinoma; Liver
Keywords: cancer; cholangiocarcinoma
MeSH Terms: conditions — Neoplasms; Cholangiocarcinoma | interventions — Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All participants (Experimental)
  Interventions: Procedure: Liver Transplantation

INTERVENTIONS:
Procedure: Liver Transplantation — Transplantation will initially be performed with deceased donor livers using the technique of caval-sparing hepatectomy unless suspected caudate involvement or caudate atrophy is a concern regarding the resection margin. Patients will be assigned a provisional Model for End-Stage Liver Disease (MELD) score by the United Network for Organ Sharing (UNOS) Regional Review Board that will make a recipient eligible for transplantation within three months at the time of listing (typically 20-24). A segment of donor iliac artery will be used as an interposition graft to the recipient infrarenal aorta. The hilus will be avoided during dissection and the bile duct, hepatic artery, and portal vein will be divided as low as possible. A frozen section of the bile duct margin will be performed and patient will undergo pancreaticoduodenectomy if positive.

SUMMARY:
Today, available therapies for hilar cholangiocarcinomas (CCA) are not satisfactory. Although these tumors are rare, their study is important because of the high death rates in afflicted patients, rivaling that of pancreatic cancer. Surgical resection offers the only current hope for long-term survival, averaging only 20% in major series1. The reality is such that for the majority of patients, CCA is a diagnosis of despair.

Although surgery has offered the only hope of cure, one of the major limiting factors in achieving long-term survival following surgical resection of CCA is the technical ability to achieve negative resection margins. The presence of malignant cells at the surgical margins following resection is a major prognostic factor predicting recurrence and death. Theoretically, the likelihood of achieving negative margins can be increased with total hepatectomy and orthotopic liver transplantation (OLT). Previous experience with OLT performed in isolation for hilar CCA's has been discouraging with dismal survival rates. However, a recent report has demonstrated that long-term survival can occur in carefully selected patients by combining the benefits of radiotherapy, chemosensitization, and OLT. With this strategy, patients survival rates of 92%, 82%, and 82% at 1, 3, and 5 years after transplantation have been achieved. It is not clear that these preliminary results can be confirmed at other centers, nor is it clear what selection criteria should optimally be used for this treatment strategy.

Our hypothesis is that select patients undergoing liver transplantation for CCA in the context of multi-modality neoadjuvant therapy exhibit survival equivalent to other established indications for liver transplantation as previously demonstrated. We will also attempt to extend previously published criteria for liver transplantation in the setting of CCA by offering this protocol to patients with evidence of intrahepatic disease and regional nodal disease. Patients undergoing transplantation for CCA will be followed longitudinally for their entire post-transplant course and compared with a matched cohort of liver transplant recipients in regard to post-transplant survival, survival on the waiting list, as well as complications pre-and post-transplantation. Explanted livers will be examined for the presence of residual tumor.

Data will be collected on the rate of regional lymph node metastasis, invasion of adjacent organs and tissues, and the rate of peritoneal metastases. The rate of tumor recurrence, site, and time to recurrence will also be assessed.

DETAILED DESCRIPTION:
Objectives Specific Aim #1: Determine whether results obtained in select patients with American Joint Commission on Cancer (AJCC) Staging System Stage I or II CCA are transferable to select patients with T3 or N1 disease.

Specific Aim #2: To determine whether success achieved with the only published protocol currently in use is directly transferable to the University of Utah's liver transplant program.

Liver Transplant Protocol:

The surgical protocol will initially be offered to liver transplant candidates with de novo hilar CCA or CCA arising in the setting of PSC. Diagnosis of CCA will be established by intraluminal brush cytology, intraluminal biopsy, or a carcinoma antigen (CA) 19.9 level greater than 100 ng / mL in the setting of a radiographic malignant stricture. Biliary aneuploidy demonstrated with DIA and FISH will be considered equivalent to cytology.

All patients with CCA will be evaluated by the liver transplant team which includes experienced hepatobiliary and liver transplant surgeons. Patients will be presented at the weekly liver transplant selection conference to assess their candidacy as well as the weekly GI Multidisciplinary Tumor Conference at the Huntsman Cancer Institute. Clinical staging prior to neoadjuvant therapy will include chest and abdominal computed tomography, liver ultrasound, and bone scan. Patients will also undergo endoscopic ultrasound with fine needle aspiration of suspicious lymph nodes. Exclusion criteria will include previous chemotherapy or radiotherapy, uncontrolled infection, a previous malignance other than non-melanoma skin cancer or in situ cervical cancer within the last five years, medical conditions precluding transplantation, metastatic disease (including N2 disease), and patients with hilar tumors extending below the cystic duct.

All patients will undergo staging laparoscopy to rule out the presence of peritoneal disease followed by staging laparotomy. Patients with extrahepatic metastases, local spread of disease to adjacent organs, and N2 nodal disease (metastasis to peripancreatic, periduodenal, periportal, celiac, superior mesenteric, and / or posterior pancreaticoduodenal nodes) will be excluded as will patients with extension of tumor into the main portal vein. Patients with N1 disease (metastasis to lymph nodes within hepatoduodenal ligament) will remain eligible for the protocol. Tumor size will not be included in the exclusion criteria. Patients with evidence of disease progression beyond study criteria will not be eligible to continue on to liver transplantation.

ELIGIBILITY:
The surgical protocol will initially be offered to liver transplant candidates with de novo hilar CCA or CCA arising in the setting of PSC. Diagnosis of CCA will be established by intraluminal brush cytology, intraluminal biopsy, or a carcinoma antigen (CA) 19.9 level greater than 100 ng / mL in the setting of a radiographic malignant stricture.

Biliary aneuploidy demonstrated with DIA and FISH will be considered equivalent to cytology.

All patients with CCA will be evaluated by the liver transplant team which includes experienced hepatobiliary and liver transplant surgeons. Patients will be presented at the weekly liver transplant selection conference to assess their candidacy as well as the weekly GI Multidisciplinary Tumor Conference at the Huntsman Cancer Institute. Clinical staging prior to neoadjuvant therapy will include chest and abdominal computed tomography, liver ultrasound, and bone scan. Patients will also undergo endoscopic ultrasound with fine needle aspiration of suspicious lymph nodes.

All patients will undergo staging laparoscopy to rule out the presence of peritoneal disease followed by staging laparotomy.

Patients with N1 disease (metastasis to lymph nodes within hepatoduodenal ligament) will remain eligible for the protocol.

Tumor size will not be included in the exclusion criteria. Patients with evidence of disease progression beyond study criteria will not be eligible to continue on to liver transplantation.

** Patients with metastatic disease are not eligible for this trial **

Exclusion criteria will include:

* previous chemotherapy or radiotherapy,
* uncontrolled infection,
* a previous malignance other than non-melanoma skin cancer or in situ cervical cancer within the last five years,
* medical conditions precluding transplantation,
* metastatic disease (including N2 disease), and
* patients with hilar tumors extending below the cystic duct.

Patients with extrahepatic metastases, local spread of disease to adjacent organs, and N2 nodal disease (metastasis to peripancreatic, periduodenal, periportal, celiac, superior mesenteric, and / or posterior pancreaticoduodenal nodes) will be excluded as will patients with extension of tumor into the main portal vein.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Schwartz, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah/Huntsman Cancer Institute, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Huntsman Cancer Institute recruited eligible participants between March 2007 and June 2011.
Groups:
- Transplant: All patients enrolled in study.
Period: Overall Study
Arm/Group | Transplant
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Transplant
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 44.8 (19.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Transplant-related Mortality
Description: Determined mortality-related transplant outcomes.
Time Frame: 2 years
Population: Entire cohort was used for analysis.
Measure: Number; unit: participants
Groups:
- Transplant: The cohort was comprised of patients who received neoadjuvant chemoradiation and transplantation.
Arm/Group | Transplant
Number analyzed (Participants) | 5
participants | 0 [0 to 52]

ADVERSE EVENTS:
Arm/Group | Transplant
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes